CLINICAL TRIAL: NCT02843126
Title: Combination of Trastuzumab and NK Immunotherapy for Recurrent Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-Trastuzumab
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Breast Cancer
Keywords: recurrent breast cancer; Her-2 positive; Trastuzumab; NK immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (2):
- Trastuzumab and NK immunotherapy (Experimental): In this group, the patients who have tumor of Her-2 positive will receive regular Trastuzumab treatment accompanied with multiple NK immunotherapy. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Trastuzumab; Biological: NK immunotherapy
- Trastuzumab (Active Comparator): In this group, the patients who have tumor of Her-2 positive will receive regular Trastuzumab to decrease tumor burden. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Pre-dose (0 hours) on Day 1 of Cycles 1 to 8 (cycle length of 21 days)
  Other Names: Herceptin
Biological: NK immunotherapy — For each procedure, 10 billion cells will be infused for 4 times
  Arms: Trastuzumab and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of Trastuzumab plus natural killer(NK) immunotherapy to recurrent breast cancer.

DETAILED DESCRIPTION:
By enrolling patients who have breast cancer of Her-2 positive adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using Trastuzumab and NK cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree evaluated by the RECIST | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Progress free survival (PFS) | 1 year
Overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Fuda cancer institute in Fuda cancer hospital, Guangzhou, Guangdong, China